CLINICAL TRIAL: NCT04996862
Title: A Study of Health Beliefs and Cancer Screening Behaviours and Intentions in Hodgkin Lymphoma Survivors
Brief Title: A Survey Exploring Health and Screening Tests in People Treated for Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp195
Record Dates: First submitted 2021-05-26; First posted 2021-08-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A survey of health beliefs and cancer screening behaviour and intentions in Hodgkin lymphoma survivors

DETAILED DESCRIPTION:
A survey of Hodgkin lymphoma survivors registered in a follow-up database, examining health beliefs (using Health Belief Model) around breast, bowel and lung cancer screening, previous screening uptake and future uptake intentions

ELIGIBILITY:
Inclusion Criteria:

* Details held in the ADAPT database at The Christie NHS Foundation trust
* Aged 18-80
* Previously treated for Hodgkin lymphoma without evidence of relapse for at least 5 years
* Treated with radiotherapy and/or alkylating agent containing chemotherapy

Exclusion Criteria:

* Have previously stated they do not wish to be contacted for research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of Hodgkin lymphoma survivors registered in a clinical follow-up database at The Christie Hospital
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
The psychosocial factors predictive of uptake of breast, bowel and lung cancer screening in HL survivors | At baseline visit
  Questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom